CLINICAL TRIAL: NCT04420468
Title: Descriptive and Retrospective Analysis of Acute Myocarditis Associated With Pandemic COVID-19 in Children
Acronym: HEART-COVID
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP200632
Record Dates: First submitted 2020-06-05; First posted 2020-06-09 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: COVID-19
Keywords: COVID-19; Acute myocarditis; Children
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Possible COVID-19 infection and acute myocarditis: Children presented with an acute myocarditis, fever and shock with a possible COVID-19 infection cared between April 2020 till the end of the main SARS-Cov-2 outbreak in 4 AP-HP Parisian hospitals :
  * Necker-Enfants Malades
  * Armand Trousseau
  * Robert Debré
  * Kremlin Bicêtre

SUMMARY:
The study objectives are to descript clinical, biological and echocardiographic features of an acute myocarditis in children in the context of COVID-19 and to identify the underlying mechanism : direct viral damage and/or inadequate host response risk.

DETAILED DESCRIPTION:
An unexpected increase of shock with fever in children suspected to be infect by the COVID-19 is observed. These children present with similar symptoms and seem to have similar clinical time course.

This unexpected phenomenon needs to be extensively described in order to further the knowledge of unusual COVID-19 presentation in children.

The study consists an extensive retrospective data collection from April 2020 till the end of the main SARS-Cov-2 outbreak, from medical file of children have exhibited acute myocarditis and cared in 4 pediatric intensive care units of Assistance Publique-Hôpitaux de Paris of Ile-de-France region.

The study objectives are to descript clinical, biological and echocardiographic features of an acute myocarditis in children in the context of COVID-19 and to identify the underlying mechanism : direct viral damage and/or inadequate host response risk.

ELIGIBILITY:
Inclusion Criteria:

* Age < 18 years
* Admitted to PICU from April 2020
* Presented with an acute myocarditis, fever and shock with a possible COVID-19 infection

Exclusion Criteria:

* Age ≥ 18 years
* Other etiologies of acute myocarditis than the COVID-19
* Opposition expressed by the holders of parental authority

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children presented with an acute myocarditis, fever and shock with a possible COVID-19 infection cared between April 2020 till the end of the main SARS-Cov-2 outbreak in 4 AP-HP Parisian hospitals :
  * Necker-Enfants Malades
  * Armand Trousseau
  * Robert Debré
  * Kremlin Bicêtre
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2020-06-10 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Acute myocarditis | 7 days
  Occurrence, description and time course of acute myocarditis
Multi-systemic inflammatory syndrome | 7 days
  Occurrence, description and time course of multi-systemic inflammatory syndrome, features of Kawasaki disease
Kawasaki disease | 7 days
  Occurrence, description and time course of features of Kawasaki disease

SECONDARY OUTCOMES:
Results of SARS-CoV-2 | 7 days
  Results of SARS-CoV-2 screening either by PCR or antibodies serological assay

CONTACTS AND LOCATIONS:
Overall Officials: Marion Grimaud, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Sylvain Renolleau, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (4):
- France (4):
  - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - Hôpital Armand Trousseau, Paris
  - Hôpital Necker-Enfants Malades, Paris
  - Hôpital Robert Debré, Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McCafferty C, Cai T, Borgel D, Lasne D, Renolleau S, Vedrenne-Cloquet M, Bonnet D, Wu J, Zaw T, Bhatnagar A, Song X, Van Den Helm S, Letunica N, Attard C, Karlaftis V, Praporski S, Ignjatovic V, Monagle P. Pathophysiological pathway differences in children who present with COVID-19 ARDS compared to COVID -19 induced MIS-C. Nat Commun. 2022 May 2;13(1):2391. doi: 10.1038/s41467-022-29951-9. PMID 35501302
- [Background] Grimaud M, Starck J, Levy M, Marais C, Chareyre J, Khraiche D, Leruez-Ville M, Quartier P, Leger PL, Geslain G, Semaan N, Moulin F, Bendavid M, Jean S, Poncelet G, Renolleau S, Oualha M. Acute myocarditis and multisystem inflammatory emerging disease following SARS-CoV-2 infection in critically ill children. Ann Intensive Care. 2020 Jun 1;10(1):69. doi: 10.1186/s13613-020-00690-8. PMID 32488505
- [Derived] Borgel D, Chocron R, Grimaud M, Philippe A, Chareyre J, Brakta C, Lasne D, Bonnet D, Toubiana J, Angoulvant F, Desvages M, Renolleau S, Smadja DM, Oualha M. Endothelial Dysfunction as a Component of Severe Acute Respiratory Syndrome Coronavirus 2-Related Multisystem Inflammatory Syndrome in Children With Shock. Crit Care Med. 2021 Nov 1;49(11):e1151-e1156. doi: 10.1097/CCM.0000000000005093. PMID 34049308